CLINICAL TRIAL: NCT00971360
Title: Proinflammatory Cytokine Levels in Patients With Conversion Disorder
Brief Title: Cytokine Levels in Conversion Disorder
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Trakya University Scientific Research Unit (TUBAB), Trakya University Scientific Research Unit (TUBAB)
Other Study IDs: TUTFEK 2009/173
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2009-09

CONDITIONS: Conversion Disorder
Keywords: conversion; cytokine; inflammation
MeSH Terms: conditions — Conversion Disorder; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conversion disorder
  Interventions: Other: conversion disorder
- Healthy control
  Interventions: Other: conversion disorder

INTERVENTIONS:
Other: conversion disorder — Proinflammatory cytokine levels in conversion disorder

SUMMARY:
The aim of this study is whether the proinflammatory cytokine levels in patients with conversion disorder is increased or not changed in the acute phase and subacute - chronic periode, compared with controls.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease

Exclusion Criteria:

* Autoimmune disease
* Neurological disease
* Any organic disorder that could possibly affect proinflammatory cytokines
* Pregnancy
* Any drug usage within 2 weeks
* Any active or passive immunization within 6 months
* Any other DSM-IV axis I psychiatric disorder
* Mental retardation
* Developmental disorder of childhood

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University Faculty of Medicine; Department of Psychiatry, Edirne, Turkey (Türkiye)

REFERENCES:
- [Background] Rief W, Pilger F, Ihle D, Bosmans E, Egyed B, Maes M. Immunological differences between patients with major depression and somatization syndrome. Psychiatry Res. 2001 Dec 31;105(3):165-74. doi: 10.1016/s0165-1781(01)00338-9. PMID 11814536
- [Background] Ziemssen T, Kern S. Psychoneuroimmunology--cross-talk between the immune and nervous systems. J Neurol. 2007 May;254 Suppl 2:II8-11. doi: 10.1007/s00415-007-2003-8. PMID 17503136
- [Background] Dantzer R. Somatization: a psychoneuroimmune perspective. Psychoneuroendocrinology. 2005 Nov;30(10):947-52. doi: 10.1016/j.psyneuen.2005.03.011. PMID 15949897